CLINICAL TRIAL: NCT02778555
Title: Development and Validation of a Daily Pain Catastrophizing Scale Based Measure
Brief Title: Development and Validation of a Daily Pain Catastrophizing Scale
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Beth Darnall, Clinical Associate Professor, Stanford University
Other Study IDs: R01AT008561-01A1 (NIH)
Record Dates: First submitted 2016-05-16; First posted 2016-05-20 (Estimated); Results first posted 2019-06-27 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Sample 1: In Sample 1 (N=186), our 14-item Daily PCS was administered daily for 14 days to replicate the 3-factor structure at the daily level, and to select the ideal 5 items for a brief Daily PCS.
  Interventions: Behavioral: Questionnaires
- Sample 2: In Sample 2 (N=209), the 5-item Daily PCS was administered daily for 14 days with short forms for PROMIS Pain Intensity, Depression, Anger, and Anxiety included on days 1, 7, and 14.
  Interventions: Behavioral: Questionnaires
- Sample 3: In Sample 3 (N=318), the 5-item Daily PCS was administered daily for 14 days with short forms for PROMIS Pain Intensity, Depression, Anger, and Anxiety included on days 1, 7, and 14. In addition, assessments of pain, mood, activity, sleep, energy level, and positive affect were administered daily for the 14-day period.
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Questionnaires

SUMMARY:
This study sought to develop and validate a brief, daily version of the Pain Catastrophizing Scale.

DETAILED DESCRIPTION:
The Pain Catastrophizing Scale (PCS; 13 items; factors: rumination, helplessness, magnification) (Sullivan 1995) measures trait catastrophizing in the context of actual or anticipated pain. Currently, there is no validated tool for measuring pain catastrophizing at the daily level. Lack of a validated daily measure stands as a barrier for studies that aim to characterize mechanisms of pain treatment and how PC adaptation / change occurs.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or above
2. Chronic pain of any etiology
3. Online access
4. Ability to participate in daily measurements over 14 days

Exclusion Criteria:

1. Lack of ability to answer questionnaires and daily catastrophizing captures, at the discretion of study staff.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with chronic pain.
Sampling Method: Non-Probability Sample
Enrollment: 713 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth D Darnall, PhD, Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Darnall BD, Sturgeon JA, Cook KF, Taub CJ, Roy A, Burns JW, Sullivan M, Mackey SC. Development and Validation of a Daily Pain Catastrophizing Scale. J Pain. 2017 Sep;18(9):1139-1149. doi: 10.1016/j.jpain.2017.05.003. Epub 2017 May 19. PMID 28528981

RESULTS

PARTICIPANT FLOW:
Groups:
- Validation Sample 1: In Sample 1 (N=186), our 14-item Daily PCS was administered daily for 14 days to replicate the 3-factor structure at the daily level, and to select the ideal 5 items for a brief Daily PCS.
- Validation Sample 2: In Sample 2 (N=209), the 5-item Daily PCS was administered daily for 14 days with short forms for PROMIS Pain Intensity, Depression, Anger, and Anxiety included on days 1, 7, and 14.
- Validation Sample 3: In Sample 3 (N=318), the 5-item Daily PCS was administered daily for 14 days with short forms for PROMIS Pain Intensity, Depression, Anger, and Anxiety included on days 1, 7, and 14. In addition, assessments of pain, mood, activity, sleep, energy level, and positive affect were administered daily for the 14-day period.
Period: Overall Study
Arm/Group | Validation Sample 1 | Validation Sample 2 | Validation Sample 3
Started | 186 | 209 | 318
Completed | 131 | 177 | 211
Not Completed | 55 | 32 | 107
Not completed — Withdrawal by Subject | 55 | 32 | 107

BASELINE CHARACTERISTICS:
Groups:
- Validation Sample 3: In Sample 3 (N=305), the 5-item Daily PCS was administered daily for 14 days with short forms for PROMIS Pain Intensity, Depression, Anger, and Anxiety included on days 1, 7, and 14. In addition, assessments of pain, mood, activity, sleep, energy level, and positive affect were administered daily for the 14-day period.
- Total: Total of all reporting groups
Arm/Group | Validation Sample 1 | Validation Sample 2 | Validation Sample 3 | Total
Number analyzed (Participants) | 131 | 177 | 211 | 519
Age, Customized [Median (Full Range); unit: years] — Measure Description: Age was collected through a categorical variable with the following categories:
  18-29; 30-39; 40-49; 50-59; 60-69; 70-79; 80+ Accordingly, median age for each sample is reported as the mean of the median range (e.g. 50-59 median range, is reported as a mean, 55) and each associated full range is listed as the median age range (e.g., 50-59).
  years
    Median Categorical Age | 55 [50 to 59] | 55 [50 to 59] | 45 [40 to 49] | 52 [18 to 100]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 122 | 186 | 417
  Male | 22 | 55 | 25 | 102

OUTCOME MEASURES:

1. Primary Outcome: Factor Analysis & PROMIS Correlation for Samples 2 & 3
Description: The validation process involves identifying, of the original 14 PCS items, which items show the largest factor loadings to the underlying factor structure that fits the data best, using model fit indices that will determine appropriate fit of the statistical model to the data, as well as convergent validity with other relevant measures (pain intensity, depression, anxiety, anger), which is tested through the use of Pearson correlations.
  Metrics used to test the hypothesis: Intraclass correlations were used to establish variability. RMSEA, CFI, TLI, and WRMR as our goodness of fit indices for arriving at 3- and 5-item measures, and to compare the measures. Reliability was tested using α. Correlations between daily pain, mood, activity, sleep, and energy were tested using pearson coefficients.
  Intent was to measure correlations between the brief PCS and the PROMIS for validation sample 2, and correlations between the brief PCS and the PROMIS for validation sample 3.
Time Frame: 14 days
Measure: Number; unit: Pearson Coefficients
Arm/Group | Validation Sample 1 | Validation Sample 2 | Validation Sample 3
Number analyzed (Participants) | 131 | 177 | 211
Pearson Coefficients
  PCS 3-item | NA — First sample, no group to correlate as PCS | .990 | NA — Not correlated with PCS 3-item as PCS 5-item was used. Primary aim for Study 3 was to correlate daily constructs (pain intensity, sleep, energy, activity, depression, anxiety, anger, positive affect)
  Pain Intensity (Daily Construct for Sample 3) | NA — First sample, no group to correlate. | .581 | .528
  Depression (Daily Construct for Sample 3) | NA — First sample, no group to correlate. | .441 | .573
  Anxiety (Daily Construct for Sample 3) | NA — First sample, no group to correlate. | .378 | .518
  Anger (Daily Construct for Sample 3) | NA — First sample, no group to correlate. | .548 | .488

ADVERSE EVENTS:
Time Frame: 9 months, 3 validation waves Adverse event data was collected during the participation period lasting 14-days. The total timeframe of study data collection was about 10 months.
Description: 9 months, 3 validation waves from the dates: 12/07/2015 to 09/21/2016
Arm/Group | Validation Sample 1 | Validation Sample 2 | Validation Sample 3
Serious Adverse Events (participants affected / at risk) | 0/186 | 0/209 | 0/318
Other Adverse Events (participants affected / at risk) | 0/186 | 0/209 | 0/318

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes